CLINICAL TRIAL: NCT06407141
Title: The Effect of Transcranial Pulse Stimulation on Cognitive Functions in Older Adults With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: The Effect of TPS on Cognitive Functions in Older Adults With MCI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEE LEUNG PONG, MSocSc Clinical Psychology Student, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSYTPS
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Arm (Experimental)
  Interventions: Behavioral: transcranial pulse stimulation
- Sham Control Arm (Sham Comparator)
  Interventions: Behavioral: Sham TMS

INTERVENTIONS:
Behavioral: transcranial pulse stimulation — Participants in the experimental arm will receive six sessions of Transcranial Pulse Stimulation (TPS) over a two-week period, using the NEUROLITH® TPS system (Storz Medical AG, Switzerland). Each session will involve delivering 6,000 ultrasound pulses at an energy level of 0.2-0.25 mJ/mm² and a frequency of 4-5 Hz, targeting specified brain regions based on MRI navigation.
  Arms: Experimental Arm
Behavioral: Sham TMS — Participants in the sham control group will undergo six sessions over a two-week period, utilizing the same NEUROLITH® TPS system (Storz Medical AG, Switzerland) as used in the experimental group. The key difference lies in the standoff device attached to the handpiece: while the experimental arm uses a standoff filled with silicone oil to transmit ultrasound pulses, the sham group's standoff is filled with air. This design ensures that the sham device replicates the appearance, feel, and sound of the active treatment without transmitting any therapeutic pulses, effectively maintaining the blinding aspect of the study.
  Arms: Sham Control Arm

SUMMARY:
The goal of this randomized controlled trial is to learn if Transcranial Pulse Stimulation (TPS) can improve cognitive functions in older adults with mild cognitive impairment (MCI). The study will also assess the safety of TPS. The main questions it aims to answer is:

Does TPS improve cognitive functions such as global cognition, attention, memory, and executive function?

Researchers will compare TPS to a sham control to evaluate the efficacy and safety of TPS in improving cognitive functions in older adults with MCI.

Participants will:

Be randomly assigned to receive either TPS or a sham intervention Undergo 6 sessions of TPS or sham intervention over a 2-week period Visit the clinic for cognitive assessments at 4 different time points (baseline, immediately post-intervention, 1-month follow-up, and 3-month follow-up) Complete questionnaires and undergo standardized neurocognitive tests, and/or MRI scans, and/or EEG assessments

The study aims to provide insights into the potential therapeutic role of TPS in enhancing cognitive functions among older adults with mild cognitive impairment.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Community-dwelling older adults aged 55 and above

Diagnosed with Mild Cognitive Impairment (MCI), classified based on:

Subjective reporting of memory deficits A score of 19-24 on the Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA) A score greater than 2 standard deviations on the Lawton Instrumental Activities of Daily Living (IADL) scale A score of 1 point or less on the AD8 questionnaire Right-handedness Ability to cooperate with assessment and intervention, without significant communicative impairments Absence of depression or anxiety, scoring less than 8 on both the Hamilton Depression Scale (HAM-D) and the Hamilton Anxiety Rating Scale (HAM-A)

Exclusion Criteria:

Current or history of dementia or other psychiatric diseases Score greater than or equal to 5 on the Hachinski Ischemic Scale (HIS) for identifying possible vascular-related causes Current or history of alcohol or drug abuse On medication within the last 2 weeks that may affect cognitive functions Report having any present neurological or psychiatric condition besides MCI Report having hemophilia, other blood clotting disorders, or medication that may cause these conditions

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Global Cognitive Function | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in global cognitive function scores from baseline, as measured by the Hong Kong version of the Montreal Cognitive Assessment (HK-MoCA). The HK-MoCA assesses various cognitive domains, including attention, memory, language, visuospatial skills, and executive functions. Scores on the HK-MoCA range from 0 to 30, with higher scores indicating better cognitive function.
Improvement in Auditory Attention | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in auditory attention scores from baseline, as measured by the Auditory Attention Span (AAS) test. This test assesses participants' ability to maintain focus on auditory stimuli and recall sequences of numbers or words. Higher scores indicate better auditory attention performance.
Improvement in Visual Attention | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in visual attention scores from baseline, as measured by the Visual Attention Span (VAS) test. The VAS test assesses the ability to maintain and recall visual stimuli. Higher scores reflect better visual attention.
Improvement in Sustained Attention | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in sustained attention scores from baseline, as measured by the Continuous Performance Test (CPT). This test evaluates sustained attention and response control, with higher scores indicating improved sustained attention over time.
Improvement in Visual-Spatial Judgment | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in visual-spatial judgment scores from baseline, as measured by the Vision Space Judgment (VSJ) test. This test evaluates the ability to judge spatial relationships between objects, with higher scores indicating improved visual-spatial judgment.
Improvement in Working Memory | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in working memory scores from baseline, as measured by the Math Problems (MP) task. This test evaluates the ability to store and manipulate information related to calculations in working memory. Higher scores indicate better working memory performance.
Improvement in Working Memory (Math) | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in working memory scores from baseline, as measured by the Math Problems (MP) task. This test evaluates the ability to store and manipulate information related to calculations in working memory. Higher scores indicate better working memory performance.
Improvement in Working Memory (General) | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in working memory scores from baseline, as measured by the Working Memory (WM) task. This test evaluates participants' ability to retain and manipulate verbal and non-verbal information. Higher scores indicate better working memory performance.
Improvement in Verbal Memory | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in verbal memory scores from baseline, as measured by the Verbal Memory List Learning (VMLL) task. This task assesses the ability to encode, store, and retrieve verbal information. Higher scores indicate improved verbal memory.
Improvement in Processing Speed | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in processing speed scores from baseline, as measured by the Symbol Digit Modality Test (SDMT). This test assesses the speed of processing visual information and converting it into a motor response. Higher scores indicate better processing speed.
Improvement in Language - Vocabulary | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in vocabulary scores from baseline, as measured by the Receptive Vocabulary (RV) task. This test evaluates participants' understanding and recognition of spoken words. Higher scores indicate improved language and vocabulary skills.
Improvement in Executive Functioning - Fluency | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in executive functioning scores from baseline, as measured by the Figural Fluency Test (FFT). This test assesses participants' ability to generate novel responses and plan effectively. Higher scores indicate better executive functioning.
Improvement in Depressive Symptoms | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in depressive symptoms from baseline, as measured by the Hamilton Depression Rating Scale (HAM-D). Higher scores indicate more severe depressive symptoms, while lower scores indicate improvement.
Improvement in Anxiety Symptoms | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in anxiety symptoms from baseline, as measured by the Hamilton Anxiety Rating Scale (HAM-A). Higher scores indicate more severe anxiety symptoms, while lower scores indicate improvement.
Improvement in Instrumental Activities of Daily Living | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in functional independence from baseline, as measured by the Hong Kong Lawton Instrumental Activities of Daily Living (IADL) Scale. Higher scores indicate greater independence in daily living activities.
Improvement in Quality of Life | Baseline, immediately post-intervention, 1-month follow-up, 3-month follow-up
  Change in quality of life scores from baseline, as measured by the Quality of Life in Alzheimer's Disease (QoL-AD) scale. Higher scores indicate better perceived quality of life.

SECONDARY OUTCOMES:
Adverse Reactions | Immediately after each TPS session
  Monitoring of adverse reactions using a self-reported questionnaire after each TPS session. The questionnaire assesses potential side effects such as headaches, dizziness, or other discomforts.

CONTACTS AND LOCATIONS:
Overall Officials: Leung Pong Lee, MOT MPsyMed, Principal Investigator — The University of Hong Kong
Locations (1):
- Department of Psychology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No